CLINICAL TRIAL: NCT01175356
Title: A COG Pilot Study of Intensive Induction Chemotherapy and 131I-MIBG Followed by Myeloablative Busulfan/Melphalan (Bu/Mel) for Newly Diagnosed High-Risk Neuroblastoma
Brief Title: Induction Therapy Including 131 I-MIBG and Chemotherapy in Treating Patients With Newly Diagnosed High-Risk Neuroblastoma Undergoing Stem Cell Transplant, Radiation Therapy, and Maintenance Therapy With Isotretinoin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANBL09P1; NCI-2011-01745 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ANBL09P1; CDR0000682629; ANBL09P1 (Other: Children's Oncology Group); ANBL09P1 (Other: CTEP); U10CA098543 (NIH); U10CA180886 (NIH)
Record Dates: First submitted 2010-08-03; First posted 2010-08-04 (Estimated); Results first posted 2017-09-28 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Ganglioneuroblastoma; Localized Resectable Neuroblastoma; Localized Unresectable Neuroblastoma; Regional Neuroblastoma; Stage 4 Neuroblastoma; Stage 4S Neuroblastoma
MeSH Terms: conditions — Ganglioneuroblastoma; Neuroblastoma | interventions — Radiotherapy, Conformal; Stem Cell Transplantation; Busulfan; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Cyclophosphamide; Doxorubicin; etoposide phosphate; Congresses as Topic; Radiation; Radiotherapy, Intensity-Modulated; 3-Iodobenzylguanidine; Isotretinoin; Melphalan; Topotecan; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (131I-MIBG, chemotherapy) (Experimental): See Detailed Description.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Procedure: Autologous Hematopoietic Stem Cell Transplantation; Drug: Busulfan; Drug: Cisplatin; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Drug: Etoposide Phosphate; Radiation: External Beam Radiation Therapy; Procedure: In Vitro-Treated Peripheral Blood Stem Cell Transplantation; Radiation: Intensity-Modulated Radiation Therapy; Radiation: Iobenguane I-131; Drug: Isotretinoin; Other: Laboratory Biomarker Analysis; Drug: Melphalan; Other: Pharmacological Study; Other: Questionnaire Administration; Procedure: Therapeutic Conventional Surgery; Drug: Topotecan Hydrochloride; Drug: Vincristine Sulfate

INTERVENTIONS:
Radiation: 3-Dimensional Conformal Radiation Therapy — Undergo radiotherapy
  Other Names: 3-dimensional radiation therapy; 3D Conformal; 3D CONFORMAL RADIATION THERAPY; 3D CRT; 3D radiotherapy; 3D-CRT; Conformal Therapy; Radiation Conformal Therapy; Radiation, 3D Conformal; Three dimensional external beam radiation therapy (procedure)
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo autologous in vitro-treated peripheral blood stem cell transplantation
  Other Names: AHSCT; Autologous; Autologous Hematopoietic Cell Transplantation; Autologous Stem Cell Transplant; Autologous Stem Cell Transplantation; Stem Cell Transplantation, Autologous
Drug: Busulfan — Given IV
  Other Names: 1, 4-Bis[methanesulfonoxy]butane; BUS; Busilvex; Bussulfam; Busulfanum; Busulfex; Busulphan; CB 2041; CB-2041; Glyzophrol; GT 41; GT-41; Joacamine; Methanesulfonic Acid Tetramethylene Ester; Methanesulfonic acid, tetramethylene ester; Mielucin; Misulban; Misulfan; Mitosan; Myeleukon; Myeloleukon; Myelosan; Mylecytan; Myleran; Sulfabutin; Tetramethylene Bis(methanesulfonate); Tetramethylene bis[methanesulfonate]; WR-19508
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; FI106; hydroxydaunorubicin; Rubex
Drug: Etoposide Phosphate — Given IV
  Other Names: Etopophos
Radiation: External Beam Radiation Therapy — Undergo radiotherapy
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiation; External Beam Radiotherapy; External Beam Radiotherapy (conventional); External Beam RT; external radiation; External Radiation Therapy; external-beam radiation; Radiation, External Beam; Teleradiotherapy; Teletherapy; Teletherapy Radiation
Procedure: In Vitro-Treated Peripheral Blood Stem Cell Transplantation — Undergo autologous in vitro-treated peripheral blood stem cell transplantation
  Other Names: in vitro-treated PBPC transplantation; in vitro-treated peripheral blood progenitor cell transplantation
Radiation: Intensity-Modulated Radiation Therapy — Undergo radiotherapy
  Other Names: IMRT; Intensity modulated radiation therapy (procedure); Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
Radiation: Iobenguane I-131 — Given IV
  Other Names: (131)I-MIBG; 131I-MIBG; I 131 Meta-iodobenzylguanidine; I-131 Metaiodobenzylguanidine; Iobenguane (131I); Iobenguane I 131; Iodine I 131 Metaiodobenzylguanidine; MIBG I-131; Raiatt MIBG-I 131
Drug: Isotretinoin — Given PO
  Other Names: 13-cis retinoic acid; 13-cis-Retinoate; 13-cis-Retinoic Acid; 13-cis-Vitamin A Acid; 13-cRA; Absorica; Accure; Accutane; Amnesteem; cis-Retinoic Acid; Cistane; Claravis; Isotretinoinum; Isotrex; Isotrexin; Myorisan; Neovitamin A; Neovitamin A Acid; Oratane; Retinoicacid-13-cis; Ro 4-3780; Ro-4-3780; Roaccutan; Roaccutane; Roacutan; Sotret; ZENATANE
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalan for Injection-Hepatic Delivery System; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813
Other: Pharmacological Study — Correlative studies
Other: Questionnaire Administration — Ancillary studies
Procedure: Therapeutic Conventional Surgery — Undergo surgery
Drug: Topotecan Hydrochloride — Given IV
  Other Names: Evotopin; Hycamptamine; Hycamtin; Nogitecan Hydrochloride; Potactasol; SKF S 104864 A; SKF S-104864-A; SKF S104864A; Topotec; Topotecan HCl; topotecan hydrochloride (oral)
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This pilot clinical trial studies induction therapy followed by iobenguane I 131 and chemotherapy in treating patients with newly diagnosed high-risk neuroblastoma undergoing stem cell transplant, radiation therapy, and maintenance therapy with isotretinoin. Radioisotope therapy, such as iobenguane I 131, releases radiation that kills tumor cells. Drugs used in chemotherapy, such as carboplatin, etoposide phosphate, busulfan, and melphalan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. A peripheral stem cell transplant may be able to replace blood-forming cells that are destroyed by iobenguane I 131 and chemotherapy. Giving radioisotope therapy, chemotherapy, and peripheral stem cell transplant may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the feasibility of treating high-risk neuroblastoma patients, age 365 days - 30 years, with a) an induction block of meta-iodobenzylguanidine labeled with iodine-131 (131I-MIBG [iobenguane I 131]) delivered after multi-agent chemotherapy, and b) post-induction busulfan/melphalan (Bu/Mel) consolidation therapy.

SECONDARY OBJECTIVES:

I. To assess the tolerability of treating high-risk neuroblastoma patients, age 365 days - 30 years, with a) an induction block of 131I-MIBG therapy delivered after multi-agent chemotherapy, and b) the tolerability of receiving post-induction Bu/Mel consolidation therapy with autologous stem-cell rescue (ASCR), and local radiation therapy.

TERTIARY OBJECTIVES:

I. To assess the response rate after a regimen of induction chemotherapy and 131I-MIBG and after a consolidation regimen of Bu/Mel with ASCR and local radiation therapy.

II. To describe the relationship of tumor norepinephrine transporter (hNET) expression with radioiodinated MIBG uptake, at diagnosis as well as with tumor response.

III. To assess the relative reliability of 123 I-MIBG and fludeoxyglucose F-18 (18FDG)-positron emission tomography (PET) imaging in assessment of tumor activity at diagnosis, and prior to surgical resection.

IV. To compare detectable tumor burden on the pre-surgical resection radioiodinated-MIBG diagnostic scan and the immediate post-MIBG therapy 131I-MIBG scan.

V. To test for the relationship of occurrence of sinusoidal obstruction syndrome (SOS) to Bu/Mel or to whole-body radiation dose or delayed radiation clearance due to 131I-MIBG.

VI. To analyze busulfan pharmacokinetics as measured by area under the curve (AUC) and relate exposure to SOS incidence.

OUTLINE:

INDUCTION CHEMOTHERAPY: Patients receive 5 courses of induction therapy.

Courses 1-2: Patients receive cyclophosphamide intravenously (IV) over 15-30 minutes and topotecan hydrochloride IV over 30 minutes on days 1-5. Patients undergo peripheral blood stem cell (PBSC) collection after course 2.

Course 3 and 5: Patients receive cisplatin IV over 1 hour on days 1-4 and etoposide phosphate IV over 1-2 hours on days 1-3. Patients undergo surgery to remove remaining tumor following course 5.

Course 4: Patients receive cyclophosphamide IV over 1-6 hours on days 1-2 and vincristine sulfate IV over 1 minute and doxorubicin hydrochloride IV over 24 hours on days 1-3.

Treatment repeats every 21 days for a total of 5 courses in the absence of disease progression or unacceptable toxicity. Patients without progressive disease proceed to iobenguane I 131 induction therapy beginning 3-6 weeks after course 5. Patients receive iobenguane I 131 IV over 90-120 minutes on day 1.

SURGERY: Patients undergo surgery after course 4 or before consolidation therapy.

CONSOLIDATION THERAPY: Within 10-12 weeks from the date of iobenguane I 131 infusion, patients receive busulfan IV over 2 hours every 6 hours on days -6 to -3 and melphalan IV on day -1.

AUTOLOGOUS STEM CELL RESCUE: Patients undergo infusion of PBSC on day 0.

RADIOTHERAPY: Beginning no sooner than 42 days after peripheral blood stem cell infusion, patients undergo 12 fractions of external-beam radiotherapy (2 dimensional [D], 3D-conformal, or intensity-modulated) to all areas of residual disease, primary tumor site, and involved nodal disease.

MAINTENANCE THERAPY: Beginning 66 days after transplantation, patients receive isotretinoin orally (PO) twice daily (BID) on days 1-14. Treatment repeats every 28 days for 6 courses.

After completion of study therapy, patients are followed up every 3 months for 1 year, every 6 months for 4 years, and then annually for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients have a diagnosis of neuroblastoma (International Classification of Diseases for Oncology [ICD-O] morphology 9500/3) or ganglioneuroblastoma verified by histology or demonstration of clumps of tumor cells in bone marrow with elevated urinary catecholamine metabolites; patients with the following disease stages at diagnosis are eligible, if they meet the other specified criteria:

  * Patients with newly diagnosed neuroblastoma with International Neuroblastoma Staging System (INSS) stage 4 are eligible with the following:

    * v-MYC myelocytomatosis viral related oncogene, neuroblastoma derived (avian) (MYCN) amplification (> 4-fold increase in MYCN signals as compared to reference signals) and age >= 365 days regardless of additional biologic features
    * Age > 18 months (> 547 days) regardless of biologic features
    * Age 12-18 months (365-547 days) with any of the following 3 unfavorable biologic features (MYCN amplification, unfavorable pathology and/or deoxyribonucleic acid [DNA] index = 1) or any biologic feature that is indeterminant/unsatisfactory/unknown
  * Patients with newly diagnosed neuroblastoma with INSS stage 3 are eligible with the following:

    * MYCN amplification (> 4-fold increase in MYCN signals as compared to reference signals), and age >= 365 days, regardless of additional biologic features
    * Age > 18 months (> 547 days) with unfavorable pathology, regardless of MYCN status
  * Patients with newly diagnosed INSS stage 2a/2b with MYCN amplification (> 4-fold increase in MYCN signals as compared to reference signals) and age >= 365 days, regardless of additional biologic features
  * Patients >= 365 days initially diagnosed with: INSS stage 1, 2, 4S who progressed to a stage 4 without interval chemotherapy; these patients must have been enrolled on ANBL00B1; it is to be noted that study enrollment must occur within 4 weeks of progression to stage 4 for INSS stage 1, 2, 4S
* Patients must have had no prior systemic therapy except for localized emergency radiation to sites of life-threatening or function-threatening disease and/or no more than 1 cycle of chemotherapy per low- or intermediate-risk neuroblastoma therapy (P9641, A3961, ANBL0531) prior to determination of MYCN amplification and histology
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 OR serum creatinine based on age and/or gender as follows:

  * =< 0.6 mg/dL (1 to < 2 years of age)
  * =< 0.8 mg/dL (2 to < 6 years of age)
  * =< 1.0 mg/dL (6 to < 10 years of age)
  * =< 1.2 mg/dL (10 to < 13 years of age)
  * =< 1.5 mg/dL (male) or 1.4 mg/dL (female) (13 to < 16 years of age)
  * =< 1.7 mg/dL (male) or 1.4 mg/dL (female) ( >= 16 years of age)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) for age
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) or serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) < 10 x ULN for age
* Shortening fraction >= 27% by echocardiogram or
* Ejection fraction >= 50% by radionuclide evaluation
* No known contraindication to peripheral blood stem cell (PBSC) collection; examples of contraindications might be a weight or size less than the collecting institution finds feasible, or a physical condition that would limit the ability of the child to undergo apheresis catheter placement (if necessary) and/or the apheresis procedure
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* Females of childbearing potential must have a negative pregnancy test; patients of childbearing potential must agree to use an effective birth control method
* Female patients who are lactating must agree to stop breast-feeding
* Patients that are 12-18 months of age with INSS stage 4 and all 3 favorable biologic features (i.e., non-amplified MYCN, favorable pathology, and DNA index > 1) are not eligible
* Patients are not eligible if they have received local radiation which includes any of the following: 1200 centigray (cGy) to more than 33% of both kidneys (patient must have at least 1 kidney that has not exceeded the dose/volume of radiation listed) or 1800 cGy to more than 30% of liver and/or 900 cGy to more than 50% of liver; emergency local irradiation is allowed prior to study entry, provided the patient still meets eligibility criteria

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 99 (Actual)
Dates: Start 2011-12-21 (Actual); Primary Completion 2016-09-28 (Actual); Study Completion 2025-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian D Weiss, Principal Investigator — Children's Oncology Group
Locations (25):
- United States (25):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Weiss BD, Yanik G, Naranjo A, Zhang FF, Fitzgerald W, Shulkin BL, Parisi MT, Russell H, Grupp S, Pater L, Mattei P, Mosse Y, Lai HA, Jarzembowski JA, Shimada H, Villablanca JG, Giller R, Bagatell R, Park JR, Matthay KK. A safety and feasibility trial of 131 I-MIBG in newly diagnosed high-risk neuroblastoma: A Children's Oncology Group study. Pediatr Blood Cancer. 2021 Oct;68(10):e29117. doi: 10.1002/pbc.29117. Epub 2021 May 24. PMID 34028986

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (131I-MIBG, Chemotherapy): Induction with multi-agent chemotherapy and MIBG labeled with iodine-131/isotretinoin/vincristine followed by Consolidation with BuMel Chemotherapy+ASCT+XRT.
Period: Overall Study
Arm/Group | Treatment (131I-MIBG, Chemotherapy)
Started | 99
Completed | 18
Not Completed | 81
Not completed — Death | 1
Not completed — Lack of Efficacy | 12
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 23
Not completed — Ineligible | 1
Not completed — Treatment Slot Not Available | 18
Not completed — Refusal by patient/parent/guardian | 6
Not completed — Pts MIBG non-avid after enrollment | 2
Not completed — On other COG study w/tumor tx intent | 7
Not completed — Inadequate stem cell for transplant | 1
Not completed — Initiation other tx prior to completion | 9

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (131I-MIBG, Chemotherapy)
Number analyzed (Participants) | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 99
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 4.2 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 86
  Unknown or Not Reported | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 18
  White | 64
  More than one race | 0
  Unknown or Not Reported | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of MIBG Avid Patients Treated With Meta-iodobenxylguanide (MIBG) Labeled With Iodine-131
Description: Number of MIBG avid patients who receive 131I-MIBG divided by the number of patients evaluable for the feasibility of MIBG endpoint x 100%.
Time Frame: Up to 6 weeks after course 5 of induction
Population: Includes patients who met criteria to receive 131I-MIBG but went off protocol therapy before receiving a dose assignment, but excludes patients that could not continue onto 131I-MIBG therapy due to lack of an open treatment slot. The definition of receiving MIBG labeled with iodine-131 is receiving 131I-MIBG.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Treatment (131I-MIBG, Chemotherapy)
Number analyzed (Participants) | 68
Percentage of participants | 86.8 [76.7 to 92.9]

2. Primary Outcome: Percentage of MIBG Avid Patients Treated With MIBG Labeled With Iodine-131 and Bu/Mel Chemotherapy
Description: Number of MIBG avid patients who receive 131I-MIBG and Bu/Mel divided by the number of patients evaluable for the feasibility of MIBG and Bu/Mel consolidation endpoint x 100%.
Time Frame: Up to day -6 of conditioning
Population: Includes patients who met criteria to receive 131I-MIBG but went off protocol therapy before receiving a dose assignment, but excludes patients that could not receive 131I-MIBG therapy due to lack of an open treatment slot. The definition of receiving Bu/Mel conditioning is receiving the first dose of planned Busulfan on Day -6 of conditioning.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Treatment (131I-MIBG, Chemotherapy)
Number analyzed (Participants) | 45
Percentage of participants | 82.2 [68.7 to 90.7]

3. Secondary Outcome: Incidence of Unacceptable Toxicity and Sinusoidal Obstruction Syndrome (SOS), Assessed by Common Terminology Criteria (CTV)v.4.0 for Toxicity Assessment and Grading for I-MIBG
Description: Number of patients who had an unacceptable toxicity or experienced SOS. Unacceptable toxicity was defined as CTC Grade 4-5 Pulmonary/Respiratory.
Time Frame: Up to 6 weeks after course 5 of induction
Population: Includes patients who received 131I-MIBG therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (131I-MIBG, Chemotherapy)
Number analyzed (Participants) | 53
Participants | 3

ADVERSE EVENTS:
Description: The Total Number of Participants at Risk (n=98) in the Adverse Events tables does not match the number of patients in the Participant Flow (n=99) because ineligible patients were excluded (n=1).
Arm/Group | Treatment (131I-MIBG, Chemotherapy)
Serious Adverse Events (participants affected / at risk) | 27/98
Other Adverse Events (participants affected / at risk) | 86/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (131I-MIBG, Chemotherapy) (N=98)
39000-Heart failure (Cardiac disorders) | 1 (1)
74500-Sinus tachycardia (Cardiac disorders) | 1 (1)
10300-Abdominal pain (Gastrointestinal disorders) | 1 (1)
14900-Ascites (Gastrointestinal disorders) | 6 (6)
55600-Mucositis oral (Gastrointestinal disorders) | 2 (2)
24600-Death NOS (General disorders) | 13 (13)
37200-General disorders and administration site conditions - Other specify (General disorders) | 1 (1)
55700-Multi-organ failure (General disorders) | 2 (2)
60600-Pain (General disorders) | 1 (1)
21600-Cholecystitis (Hepatobiliary disorders) | 1 (1)
40000-Hepatic failure (Hepatobiliary disorders) | 2 (2)
40400-Hepatic pain (Hepatobiliary disorders) | 2 (2)
40600-Hepatobiliary disorders - Other specify (Hepatobiliary disorders) | 2 (2)
66500-Portal hypertension (Hepatobiliary disorders) | 3 (3)
44800-Infections and infestations - Other specify (Infections and infestations) | 2 (2)
53100-Lung infection (Infections and infestations) | 1 (1)
73700-Sepsis (Infections and infestations) | 3 (3)
10900-Activated partial thromboplastin time prolonged (Investigations) | 2 (2)
11600-Alanine aminotransferase increased (Investigations) | 4 (4)
15000-Aspartate aminotransferase increased (Investigations) | 4 (4)
17400-Blood bilirubin increased (Investigations) | 8 (8)
45800-INR increased (Investigations) | 2 (2)
88200-Weight gain (Investigations) | 5 (5)
88300-Weight loss (Investigations) | 2 (2)
10700-Acidosis (Metabolism and nutrition disorders) | 1 (1)
13500-Anorexia (Metabolism and nutrition disorders) | 1 (1)
41600-Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
41800-Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
42600-Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
43100-Hypokalemia (Metabolism and nutrition disorders) | 2 (3)
43300-Hyponatremia (Metabolism and nutrition disorders) | 3 (3)
58000-Neoplasms benign malignant and unspecified (incl cysts and polyps) - Other specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
72500-Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1 (1)
43900-Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (5)
65900-Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
69000-Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
71600-Respiratory thoracic and mediastinal disorders - Other specify (Respiratory, thoracic and mediastinal disorders) | 1 (1)
43600-Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (131I-MIBG, Chemotherapy) (N=98)
13200-Anemia (Blood and lymphatic system disorders) | 24 (49)
33300-Febrile neutropenia (Blood and lymphatic system disorders) | 54 (81)
20000-Cardiac arrest (Cardiac disorders) | 1 (1)
78900-Supraventricular tachycardia (Cardiac disorders) | 1 (1)
38900-Hearing impaired (Ear and labyrinth disorders) | 9 (11)
10100-Abdominal distension (Gastrointestinal disorders) | 1 (1)
10300-Abdominal pain (Gastrointestinal disorders) | 7 (7)
14900-Ascites (Gastrointestinal disorders) | 5 (5)
22100-Colitis (Gastrointestinal disorders) | 1 (1)
25700-Diarrhea (Gastrointestinal disorders) | 6 (7)
29400-Enterocolitis (Gastrointestinal disorders) | 1 (1)
36400-Gastritis (Gastrointestinal disorders) | 1 (1)
44600-Ileus (Gastrointestinal disorders) | 1 (1)
55600-Mucositis oral (Gastrointestinal disorders) | 19 (22)
57600-Nausea (Gastrointestinal disorders) | 15 (17)
59700-Oral pain (Gastrointestinal disorders) | 2 (2)
81900-Typhlitis (Gastrointestinal disorders) | 1 (1)
87900-Vomiting (Gastrointestinal disorders) | 18 (20)
33900-Fever (General disorders) | 1 (1)
37200-General disorders and administration site conditions - Other specify (General disorders) | 1 (1)
60600-Pain (General disorders) | 7 (8)
12000-Allergic reaction (Immune system disorders) | 1 (1)
13100-Anaphylaxis (Immune system disorders) | 1 (1)
20500-Catheter related infection (Infections and infestations) | 10 (11)
25600-Device related infection (Infections and infestations) | 1 (1)
44800-Infections and infestations - Other specify (Infections and infestations) | 17 (18)
53100-Lung infection (Infections and infestations) | 2 (2)
61100-Pancreas infection (Infections and infestations) | 1 (1)
73700-Sepsis (Infections and infestations) | 4 (4)
74600-Sinusitis (Infections and infestations) | 1 (1)
75200-Skin infection (Infections and infestations) | 1 (1)
76000-Small intestine infection (Infections and infestations) | 1 (1)
82300-Upper respiratory infection (Infections and infestations) | 1 (1)
83100-Urinary tract infection (Infections and infestations) | 4 (4)
88900-Wound infection (Infections and infestations) | 2 (2)
13800-Aortic injury (Injury, poisoning and procedural complications) | 1 (1)
45700-Injury poisoning and procedural complications - Other specify (Injury, poisoning and procedural complications) | 1 (1)
47300-Intraoperative hepatobiliary injury (Injury, poisoning and procedural complications) | 1 (1)
47700-Intraoperative renal injury (Injury, poisoning and procedural complications) | 1 (1)
10900-Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
11600-Alanine aminotransferase increased (Investigations) | 14 (15)
15000-Aspartate aminotransferase increased (Investigations) | 14 (14)
17400-Blood bilirubin increased (Investigations) | 1 (1)
24100-Creatinine increased (Investigations) | 2 (2)
34000-Fibrinogen decreased (Investigations) | 1 (1)
37500-GGT increased (Investigations) | 1 (1)
52600-Lipase increased (Investigations) | 1 (1)
53700-Lymphocyte count decreased (Investigations) | 21 (49)
58300-Neutrophil count decreased (Investigations) | 27 (56)
65800-Platelet count decreased (Investigations) | 28 (59)
88200-Weight gain (Investigations) | 1 (1)
88300-Weight loss (Investigations) | 1 (1)
88500-White blood cell decreased (Investigations) | 23 (50)
10700-Acidosis (Metabolism and nutrition disorders) | 1 (1)
13500-Anorexia (Metabolism and nutrition disorders) | 33 (48)
24700-Dehydration (Metabolism and nutrition disorders) | 12 (12)
41300-Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
41400-Hyperglycemia (Metabolism and nutrition disorders) | 9 (12)
41600-Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
41700-Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
41800-Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
42600-Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3)
42700-Hypocalcemia (Metabolism and nutrition disorders) | 3 (3)
42900-Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
43100-Hypokalemia (Metabolism and nutrition disorders) | 33 (36)
43200-Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
43300-Hyponatremia (Metabolism and nutrition disorders) | 8 (9)
43500-Hypophosphatemia (Metabolism and nutrition disorders) | 16 (18)
54900-Metabolism and nutrition disorders - Other specify (Metabolism and nutrition disorders) | 2 (2)
18200-Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
37300-Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
60700-Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
10500-Abducens nerve disorder (Nervous system disorders) | 1 (1)
38800-Headache (Nervous system disorders) | 2 (2)
79100-Syncope (Nervous system disorders) | 1 (1)
11400-Agitation (Psychiatric disorders) | 2 (2)
13700-Anxiety (Psychiatric disorders) | 1 (1)
25400-Depression (Psychiatric disorders) | 1 (1)
11100-Acute kidney injury (Renal and urinary disorders) | 1 (1)
39300-Hematuria (Renal and urinary disorders) | 2 (2)
71100-Renal calculi (Renal and urinary disorders) | 1 (1)
19300-Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
29700-Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (4)
43900-Hypoxia (Respiratory, thoracic and mediastinal disorders) | 8 (8)
64900-Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
66400-Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
68700-Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
69000-Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
71500-Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
78100-Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (2)
74700-Skin and subcutaneous tissue disorders - Other specify (Skin and subcutaneous tissue disorders) | 1 (1)
79000-Surgical and medical procedures - Other specify (Surgical and medical procedures) | 1 (1)
39100-Hematoma (Vascular disorders) | 1 (1)
42100-Hypertension (Vascular disorders) | 1 (2)
43600-Hypotension (Vascular disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior approval.